CLINICAL TRIAL: NCT03770338
Title: Effect of 1 Month Preoperative Teriparatide Use on the Insertional Torque of Pedicle Screws for Lumbar Fusion Surgery
Brief Title: Preoperative Teriparatide Use on Insertional Torque of Pedicle Screws for Lumbar Fusion Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Teriparatide_RCT
Record Dates: First submitted 2018-12-03; First posted 2018-12-10 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Osteoporosis; Fusion of Spine, Lumbar Region
Keywords: osteoporosis, teriparatide, insertional torque
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Intervention Model Description: To detect any significant difference between control and teriparatide groups in terms of intraoperative insertional torque strength
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Recruitment for fusion surgery as usual
- Teriparatide (Experimental): Preoperative 1 month use of teriparatide, before lumbar fusion surgery
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — 20ug dosage daily injection, 1-month preoperative
  Other Names: Forteo
  Arms: Teriparatide

SUMMARY:
This project aims to investigate any difference of insertional torque strength for osteoporotic patients with preoperative 1-month teriparatide injections versus those without. The increased insertional torque of pedicle screws during surgery after only 1 month of teriparatide use has also been studied. However, the effect of teriparatide on vertebral body bone mineral density (BMD) prior to and after fusion surgery has not been studied. The effects on screw insertional torque has also not been studied via a randomized controlled trial method.

DETAILED DESCRIPTION:
For this project, adult patients (>40 years) undergoing lumbar spinal fusion will be randomized to undergo teriparatide treatment for 1 month prior to surgery. Patients will have their baseline BMD assessed by DEXA scan must be considered as osteoporotic (>2.5 SD from sex-matched young adult, or previous vertebral and/or femoral fractures) and indicated for spinal fusion surgery to undergo study. Exclusion criteria included Paget disease of bone, high laboratory tests for serum alkaline phosphatase or calcium, previous radiation treatment or fusion surgery to lumbar spine, bone tumors, metabolic bone disease, and hypersensitivity to teriparatide. Surgery involving single- or multi-level lumbar spinal fusion for any of the conditions: lumbar spinal stenosis, degenerative/isthmic/congenital spondylolisthesis, degenerative scoliosis. Only the surgeon and assessors will be blinded as patients will know their treatment arm.

Patients undergo a quantitative CT prior to initiation of teriparatide treatment. After one month of Teriparatide treatment, the drug is discontinued with another DEXA scan to see the changes in BMD. A quantitative CT will be performed after surgery and at 6 months postoperatively. Follow-up schedules include preoperative, immediate postoperative, postoperative 6 weeks, 3 months, 6 months, 12 months and at 24 months. At all follow-up timepoints, any complications, fusion demonstrated by cross-trabeculation on x-rays (with final confirmation at the 6 month CT), and objective questionnaires for quality of life including the EuroQoL 5 dimensions 5-level questionnaire (EQ-5D-5L), back pain numeric rating scale (NRS), osteoporosis assessment questionnaire-physical function (OPAQ-PF) and ambulatory status assessment (ASA) questionnaires will be recorded. Other quality-of-life scores include ODI and SF-36, along with adherence evaluation of osteoporosis treatment (ADEOS), osteoporosis attitude questionnaire and osteoporosis knowledge questionnaire. Once a patient is identified to be suitable for this protocol, they will need to be assessed by a medical social worker to be unable to afford this entire treatment regimen before institutional support for the drug treatment is provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be osteoporotic: baseline BMD assessed by DEXA scan must be considered as osteoporotic (>2.5 SD from sex-matched young adult, or previous vertebral and/or femoral fractures) and indicated for spinal fusion surgery

Exclusion Criteria:

* Paget disease of bone, high laboratory tests for serum alkaline phosphatase or calcium, previous radiation treatment or fusion surgery to lumbar spine, bone tumors, metabolic bone disease, and hypersensitivity to teriparatide

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Insertional torque Intraoperative insertional torque measurement | Intraoperative
  Measurement of the insertional torque of pedicle screws

SECONDARY OUTCOMES:
Bone Mineral Density (BMD) | Preoperative, Immediate postop and 6 month postop dual energy x-ray absorptiometry (DEXA) scan
  Assessment of BMD before and after treatment
Complication rate | Baseline, immediate postop, postop 6 weeks, postop 3 months, postop 6 months, postop 12 months, postop 24 months
  screw loosening, fracture, non-union
Fusion rate | At 6 months CT
  Fusion rate assessment
EQ-5D-5L | Baseline, immediate, postop 6 weeks, postop 3 months, postop 6 months, postop 12 months, postop 24 months
  Utility score
Oswestry Disability Index (ODI) | Baseline, immediate postop, postop 6 weeks, postop 3 months, postop 6 months, postop 12 months, postop 24 months
  Assessment of disability
Short form 36-item questionnaire (SF-36) | Baseline, immediate postop, postop 6 weeks, postop 3 months, postop 6 months, postop 12 months, postop 24 months
  General quality of life score
Numeric Rating Scale (NRS) | Baseline, immediate postop, postop 6 weeks, postop 3 months, postop 6 months, postop 12 months, postop 24 months
  This is a self-perceived severity of back pain. The scores range from minimum 0 (no pain) to maximum 10 (most painful) in a scale of severity. Hence, a higher value represents worse outcome. There are two subquestions: 1) What the patient indicates as the most severe pain in the past 24 hours of answering the questionnaire; 2) The patient indicates the score of the usual pain status in the past 24 hours. 0 represents no pain, 1-3 represents mild pain (nagging, annoying, interfering little with ADLs), 4-6 represents moderate pain (interferes significantly with ADLs), and 7-10 represents severe pain (disabling; unable to perform ADLs).
Osteoporosis Assessment Questionnaire-Physical Function (OPAQ-PF) | Baseline, immediate postop, postop 6 weeks, postop 3 months, postop 6 months, postop 12 months, postop 24 months
  This is a general osteoporosis score with 15 questions split into three categories (mobility, balance and transfer). A Likert scale of 6 answers are possible for each question from "no difficulties" to "unable to perform" in a scale of severity. A total score can be tabulated from adding all domain scores. Higher values indicate better outcome. A 0-100 scale provides a total score, where 0 indicates the worst health status and 100 no difficulties.
Ambulatory status assessment (ASA) | Baseline, immediate postop, postop 6 weeks, postop 3 months, postop 6 months, postop 12 months, postop 24 months
  Functional assessment
Adherence evaluation of osteoporosis treatment (ADEOS) | Baseline, immediate postop, postop 6 weeks, postop 3 months, postop 6 months, postop 12 months, postop 24 months
  Osteoporosis treatment assessment
Osteoporosis attitude and knowledge questionnaire | Baseline, immediate postop, postop 6 weeks, postop 3 months, postop 6 months, postop 12 months, postop 24 months
  To assess patients' understanding of the disease and their views towards osteoporosis

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (3):
  - Jason Pui Yin Cheung, Hong Kong, Please Select An Option Below
  - Duchess of Kent Children's Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong